CLINICAL TRIAL: NCT05093816
Title: An Online Wellness Intervention for University Students: Investigating the Efficacy of The Common Elements Toolbox in the UK
Brief Title: Evaluating a Single-session Mental Health Intervention for UK University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-212
Record Dates: First submitted 2021-10-01; First posted 2021-10-26 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Depression; Anxiety; Happiness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Tooplbox (Experimental)
  Interventions: Behavioral: Common Elements Toolbox
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: Common Elements Toolbox — The Common Elements Toolbox (COMET) is an online single-session intervention. It is entirely self-guided and lasts about 60 minutes. Participants complete a series of reading and writing exercises focused on four modules: cognitive restructuring, behavioral activation, gratitude, and self-compassion. The intervention is entirely unguided and completed in a single sitting.
  Arms: Common Elements Tooplbox

SUMMARY:
The investigators are evaluating if an online single-session intervention, the Common Elements Toolbox (COMET) can improve mental health and wellbeing among UK university students.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to four weeks post-intervention
  Measure of depressive symptoms. Scores range from 0-27, with higher scores indicating greater levels of depression.
Generalized Anxiety Disorder 7-item Checklist (GAD-7) | Change from baseline to four weeks post-intervention
  Measure of anxiety symptoms. Scores range from 0-21, with higher scores indicating greater levels of anxiety.
Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). | Change from baseline to four weeks post-intervention
  Measure of wellbeing. Scores range from 7-35, with higher scores indicating greater well-being.
Positive and Negative Affect Schedule | Change from baseline to four weeks post-intervention
  A measure of positive affect and negative affect. Scores on the positive affect subscale range from 10-50, with higher scores indicating greater positive affect. The negative affect subscale also ranges from 10-50, with greater scores indicating greater levels of negative affect.
Acceptability of Intervention Measure (AIM) | Post-intervention (immediately after participants complete the intervention)
  Measure of acceptability. Scores range from 4-20, with higher scores indicating greater acceptability.
Intervention Appropriateness Measure | Post-intervention (immediately after participants complete the intervention)
  Measure of appropriateness. Scores range from 4-20, with higher scores indicating greater appropriateness.

IPD SHARING:
Plan to Share IPD: Undecided